CLINICAL TRIAL: NCT06875648
Title: Intestinal Flora Differences Between Colorectal Cancer Patients and Healthy Individuals: A Case-Control Study
Brief Title: Intestinal Flora Differences Between Colorectal Cancer Patients and Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Hansung University (Other)
Responsible Party: Sponsor
Other Study IDs: GDMEC-2024-028
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Gut Microbiota Dysbiosis
Keywords: Colorectal Neoplasms (MeSH); Gastrointestinal Microbiome (MeSH); Dysbiosis (MeSH); Microbial Biomarkers
MeSH Terms: conditions — Colorectal Neoplasms; Dysbiosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biospecimen Type: Fecal samples (preserved for microbial DNA analysis). Collection: Collected retrospectively from colorectal cancer (CRC) patients at diagnosis and healthy controls during routine check-ups.
  Storage: Archived at -80°C in hospital biobanks prior to DNA extraction.
  Processing:
  DNA extracted from fecal samples using standardized kits (e.g., QIAamp DNA Stool Mini Kit).
  Focus on bacterial genomic DNA (e.g., 16S rRNA gene sequencing targeting V3-V4 regions or whole-genome shotgun metagenomics).
  Quality Control: DNA concentration and purity verified via spectrophotometry (e.g., NanoDrop) and gel electrophoresis.
  Purpose: To characterize gut microbiota composition (bacterial taxa abundance) and compare CRC patients vs. healthy controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRC Patients: Participants: 36 individuals with histopathologically confirmed colorectal cancer.
  Data Source: Archived fecal samples and medical records from patients diagnosed between January 2022 and October 2023.
  Inclusion Criteria:
  Adults (≥18 years). Newly diagnosed CRC without prior chemotherapy/radiotherapy. Availability of fecal samples collected at diagnosis.
  Exclusion Criteria:
  Antibiotic/probiotic use within 3 months before sample collection. Concurrent gastrointestinal infections or inflammatory bowel disease. Subgroups: Stratified by clinical stage (I, II, III) based on TNM classification from medical records.
  Interventions: Other: Not applicable (observational study)
- Healthy Controls: Participants: 25 age- and gender-matched individuals without gastrointestinal diseases or cancer history.
  Data Source: Archived fecal samples and health screening records from routine check-ups during the same period.
  Inclusion Criteria:
  Adults (≥18 years). No history of colorectal polyps, cancer, or chronic gastrointestinal disorders. Normal colonoscopy or fecal occult blood test results.
  Exclusion Criteria:
  Antibiotic/probiotic use within 3 months before sample collection. Recent acute gastrointestinal symptoms (e.g., diarrhea, constipation).
  Interventions: Other: Not applicable (observational study)

INTERVENTIONS:
Other: Not applicable (observational study) — Retrospective analysis of gut microbiota in CRC patients vs. healthy controls. No interventions were administered; data were collected from archived samples and medical records.

SUMMARY:
This observational case-control study aims to compare the composition of intestinal microbiota between colorectal cancer (CRC) patients and healthy individuals. Fecal samples from 36 CRC patients and 25 healthy controls were analyzed for bacterial abundance. Results indicate significant differences in beneficial, neutral, and harmful bacterial populations between groups, with CRC patients showing reduced beneficial flora (e.g., Lactobacillus) and increased harmful/neutral flora (e.g., Staphylococcus). Further stratification by cancer stage (I-III) revealed progressive dysbiosis with disease progression.

DETAILED DESCRIPTION:
This observational case-control study investigates the compositional differences in intestinal microbiota between individuals diagnosed with colorectal cancer (CRC) and healthy controls. The study enrolled 36 CRC patients confirmed by histopathology and 25 age- and gender-matched healthy volunteers without gastrointestinal diseases or antibiotic/probiotic use within the preceding three months. Fecal samples were collected from CRC patients at the time of diagnosis and from healthy participants during routine health screenings. Utilizing 16S rRNA sequencing or quantitative PCR, the relative abundance of specific bacterial taxa (e.g., Lactobacillus, Bifidobacterium, Staphylococcus) was quantified to assess dysbiosis patterns. Additionally, the analysis stratified CRC patients by clinical stage (I-III) to explore progressive shifts in microbial communities with disease advancement. The findings aim to elucidate the role of gut microbiota in CRC pathogenesis and provide insights into potential microbiome-based diagnostic or therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with histopathologically confirmed colorectal cancer (CRC group)
* Archived fecal sample available from time of CRC diagnosis (prior to treatment)
* Complete clinical records including TNM staging (I-III) for CRC patients
* Age- and gender-matched adults without CRC history (control group)
* Archived fecal sample available from routine health check-ups (control group)

Exclusion Criteria:

* Recent antibiotic or probiotic use (within 3 months)
* History of inflammatory bowel disease
* Incomplete medical records
* For controls: history of colorectal cancer, polyps, or chronic gastrointestinal diseases
* For controls: abnormal colonoscopy or fecal occult blood test within the past year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective case-control study of 36 CRC patients (stages I-III, diagnosed 2022-2023) and 25 healthy controls from Central Hospital, Zhanjiang, China. CRC group: pre-treatment fecal samples, TNM staging. Control group: age/gender-matched, no GI diseases, normal colonoscopy/fecal tests. Exclusions: antibiotic/probiotic use (past 3 months), inflammatory bowel disease, incomplete records.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Mean Relative Abundance of Intestinal Bacterial Genera between CRC Patients and Healthy Controls | Retrospective analysis of fecal samples collected between January 2021 and March 2025
  The primary metric is the mean relative abundance of specific intestinal bacterial genera (e.g., Lactobacillus, Bifidobacterium, Staphylococcus). Quantitative comparison will be performed between CRC patients and healthy controls using data obtained from fecal samples via 16S rRNA sequencing or qPCR. This is a retrospective analysis of samples collected between January 2021 and March 2025.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital of Guangdong Provincial Nongken, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to restrictions imposed by the hospital ethics committee and Chinese data privacy laws.